CLINICAL TRIAL: NCT03805828
Title: The Effectiveness of an Educational Program on Parenting Stress and Coping Mechanism Among Parents of Children With Autism Spectrum Disorder in Amman, Jordan
Brief Title: Effectiveness of Educational Program on Parenting Stress and Coping Mechanism Among Parents of Children With Autism Spectrum Disorder in Amman, Jordan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Haytham Mohammad Al-Oran, principle investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University Putra Malaysia
Record Dates: First submitted 2019-01-08; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism spectrum disorder; parenting stress; coping mechanism; coping strategies; education program; educational intervention
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expermental (Experimental): In the intervention group, the educational program will deliver as a one-day event in four sessions: (1)background of autism spectrum disorder(ASD) and coping mechanism,(2) targeting communication and social difficulties among ASD children using coping mechanism,(3) targeting behavior problems among ASD children using coping mechanism, and (4) stress management as coping mechanism.
  Interventions: Other: Educational program on parenting stress and coping mechanism
- Control (Active Comparator): In the control group, the educational about communicable disease among childhood deliver as a one-day event in four sessions: (1) introduction and background communicable disease of childhood,(2) communicable diseases of childhood (Chicken Pox, Diphtheria,and pertussis[a whooping cough]),(3) communicable diseases of childhood (Measles,Mumps,rubella[German Measles]and Poliomyelitis(,and (4) infection control.
  Interventions: Other: Educational program on parenting stress and coping mechanism

INTERVENTIONS:
Other: Educational program on parenting stress and coping mechanism — The educational program will deliver as a one-day event in four sessions: (1)background of autism spectrum disorder(ASD) and coping mechanism,(2) targeting communication and social difficulties among ASD children using coping mechanism,(3) targeting behavior problems among ASD children using coping mechanism, and (4) stress management as coping mechanism. The contents of the educational program deliver through the use of PowerPoint slides, Whiteboard and marker, practical exercise, video clips followed by group discussion and provision a hard copy booklet containing all items which were supposed to discuss. As well as each session will approximately be taken one hour. Each group will consist of 10 participants.

SUMMARY:
Health and well being of children are inextricably linked to the physical, emotional and psychological of their parents. Autism Spectrum Disorder is one of the neurological developmental disorders characterized by moderate to severe impairments in social interactions, language, and cognitive development, as well as included repetitive behaviors, restricted interests, and emotional distress. Coping with a stressful situation is classified as one of the most challenges in one's life. The overall aim of this study is to examine the effectiveness of the educational program on parenting stress and coping mechanism among parents of children with ASD in Amman, Jordan at baseline, post-test and at two months follow-up assessment. Two hundred parents of children with Autism spectrum disorder will be assigned to the intervention group (n = 100) and the control group (n = 100). Measures of parent stress and coping mechanism using the parent stress index(PSI) and Brief COPE will administer at pre-, post-treatment, and 2-months follow-up.

DETAILED DESCRIPTION:
Background: Health and well being of children are inextricably linked to the physical, emotional and psychological of their parents. Maintaining the health and well-being of parents is a precondition for the best optimal care of their children with Autism Spectrum Disorder (ASD). The overall aim of the current study is to evaluate the effectiveness of an educational program on parenting stress and coping mechanism among parents of children with ASD in Jordan.

Methods: A cluster randomized controlled trial will be conducted in 4 private centers for the treatment of Autistic Disorder in Amman, Jordan. Inclusion criteria: father or mother of a child who diagnosed for the period of three years since the initial time of diagnosis, father or mother who provides care and living together with the child, father or mother has the ability to read and write Arabic, father or mother age above 20 years old,and center provides caring just for ASD child with age 12 years and younger. Exclusion criteria: father or mother whose child had other chronic or illnesses (e.g, type 1 diabetes, down syndrome, learning disabilities, fetal alcohol syndrome), foreign father or mother of a child with ASD residents in Amman, father or mother who previously participated in the intervention research (e.g, Cognitive Behavior Therapy, Mindfulness-Based Intervention), father or mother of a child who takes any pharmacologic management of ASD (e.g,Risperdal, Ritalin), father or mother with more than one child diagnosed with ASD,and center doesn't include a suitable classroom for implementing the intervention program. The educational intervention program will deliver to the intervention group as a one-day event in four sessions. Whereas, the control group will receive education about the communicable disease among childhood. With an estimated effect design of 1.3, a cluster size of 4 and 20% non-completion, the trial will need to enroll 200 participants. The primary outcomes of the current study are parenting stress and coping mechanism scores, which will be assessed using the Parent Stress Index-Short Form and Brief COPE, respectively. parenting stress and coping mechanism scores will be assessed at pre-intervention, post-intervention and follow-ups at week 8.

Results: The parenting stress and the coping mechanism will be compared between the intervention and control groups using A 2×3 repeated measure ANOVA.

Conclusions: Hypothesize that primary outcomes will improve significantly after the intervention compared to the control group. The finding from this study will determine the effectiveness of the educational program on parenting stress and coping mechanism among Jordanian parents of children with ASD. If proven to be effective, the educational program can serve as a part of therapeutic plan support to reduce parenting stress and improve coping mechanism.

ELIGIBILITY:
Inclusion Criteria:

The participant's inclusion eligibility criteria:

* Father or mother of a child who diagnosed for the period of three years since the initial time of diagnosis
* Father or mother who provides care and living together with the child
* Father or mother has the ability to read and write Arabic, and (4) father or mother age above 20 years old

The center's inclusion eligibility criteria:

* Center provides caring only for ASD child with age 12 years and younger
* Provide the following services: speech, language, occupational, physiotherapy, educational, nutrition and medical services.

Exclusion Criteria:

The participant's exclusion eligibility criteria

* Father or mother whose child had other chronic or illnesses (e.g, type 1 diabetes, down syndrome, learning disabilities, fetal alcohol syndrome)
* Foreign father or mother of a child with ASD residents in Amman
* Father or mother who previously participated in the intervention research (e.g, Cognitive Behavior Therapy, Mindfulness-Based Intervention)
* Father or mother of a child who takes any pharmacologic management of ASD (e.g,Risperdal, Ritalin)
* Father or mother with more than one child diagnosed with ASD

The center's exclusion eligibility criteria

* Center doesn't include a suitable classroom for implementing the intervention program

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
parenting stress | Mean change in scores of parenting stress from baseline to endpoint(two months follow-up) assessment
  Self reported 36 statements on three subscales: parental distress (PD), parent-child dysfunctional interaction (P-CDI), and difficulty of the child (DC). Each subscale contains 12 items. The PSI-SF rated on a 5-point Likert scale, include 1 (strongly disagree) , 2 ( disagree ), 3 ( not sure ), 4 (agree) 5 (strongly agree), total scores range from 36 to 180. On the PSI-SF, stress levels considered normal with less than 90 scores , whereas , high-stress considered at or above the 90 scores
coping mechanism | Mean change in scores of coping mechanism from baseline to endpoint(two months follow-up) assessment
  self-administered questionnaire twenty-eight items of the Brief COPE are grouped into fourteen subscales containing two items for each: acceptance, active coping, planning, behavioral disengagement, denial, substance use, humor, positive reframing, religious coping, self-blame, self-distraction, use of emotional support, use of instrumental support, and venting emotions . The items of subscale rated on a four-point Likert scale with a response for each item ranging from 1 ( I haven't been doing this at all ) to 4 (I have been doing this a lot)

CONTACTS AND LOCATIONS:
Locations (2):
- Jordan (2):
  - Centers for the treatment of Autistic Disorder, Amman
  - Ministry of Social Development, Amman

IPD SHARING:
Plan to Share IPD: Yes
Primary outcomes measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within 7 months
Access Criteria: Date request will be reviewed by an external independent review panel. Requesters will be required to sign the data access agreement